CLINICAL TRIAL: NCT06432881
Title: Investigation of Skin Pigmentation Effect on Performance of Masimo Pulse Oximetry (INSPIRE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GOOD0001
Record Dates: First submitted 2024-02-23; First posted 2024-05-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-10

CONDITIONS: Hypoxemia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- RD SET Sensor (Experimental): All subjects are enrolled into this arm and will have Sp02 measurements obtained.
  Interventions: Device: RD SET Sensor

INTERVENTIONS:
Device: RD SET Sensor — All subjects are enrolled into this arm and will have Sp02 measurements obtained.

SUMMARY:
The objective of this study is to evaluate the performance of Masimo RD SET® SpO2 sensors in subjects with light and dark skin pigmentation in the intensive care therapeutic area.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older.
* Subject is receiving care in an intensive care unit.
* Subject with an arterial catheter in place.
* Subject is experiencing hypoxemia as defined by 1) need for supplement oxygen or 2) peripheral oxygenation ≤ 94% on room air

Exclusion Criteria:

* Subjects in whom pulse oximetry cannot be reliably performed on both the third and fourth digit on the hand ipsilateral to the arterial line, precluding application of the sensor (e.g., amputation and deformity).
* Subjects with a skin condition affecting the digits, where the sensor is applied, which would preclude sensor placement as standard of care (e.g., psoriasis, eczema, angioma, scar tissue, burn, fungal infection, substantial skin breakdown, etc.).
* Subjects with distinct geographic variances in skin pigmentation (e.g., vitiligo) on the digit where the sensor is applied, which would preclude sensor placement as standard of care.
* Subjects with nail polish or acrylic nails on the digits where sensor needs to be applied.
* Subjects with known allergic reactions to adhesive tapes.
* Subjects with arterial catheter placed in a lower extremity.
* Subjects not suitable for the investigation at the discretion of the investigator or the clinical team.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Investigation of skin pigmentation effect on performance of Masimo pulse oximetry | Approximately 30 minutes
  The study is designed to evaluate the performance of Masimo RD SET SpO2 sensors in subjects with light and dark skin pigmentation in the intensive care therapeutic area. SpO2 accuracy will be determined by calculating the ARMS value which will be reported as percent of oxygen saturated hemoglobin.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States